CLINICAL TRIAL: NCT06887998
Title: The Effect of Two Different Doses of Oral Gabapentin on Sevoflurane-associated Emergence Agitation and Delirium in Adult Patients After Nasal Surgery. A Prospective Controlled, Randomized, Double-blinded Study.
Brief Title: The Effect of Oral Gabapentin on Emergence Agitation and Delirium in Adult Patients After Nasal Surgery.
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Maged Mobarak Abdelkhalek Abdelfattah, assisstant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: gabapentin for agitation
Record Dates: First submitted 2025-02-02; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-02

CONDITIONS: Emergence Agitation
Keywords: emergence agitation; gabapentin; nasal surgery
MeSH Terms: conditions — Emergence Delirium | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Patients will be randomly allocated (using sealed opaque numbered envelopes indicating the group of each patient, carried out by an independent anesthesiologist) into one of three groups :
  * Group (A) [n = 21 patients]: will receive 600 mg oral gabapentin one hour before induction.
  * Group(B) [n =21 patients ]:will receive 400 mg oral gabapentin one hour before induction.
  * Group (C) (control group) [n =21 patients ] : will receive placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Gabapentin 600 mg group (Active Comparator): 21 patients will receive 600 mg oral gabapentin one hour before induction.
  Interventions: Drug: Gabapentin 600 mg capsules
- Gabapentin 400 mg group (Active Comparator): 21 patients will receive 400 mg oral gabapentin one hour before induction.
  Interventions: Drug: Gabapentin 400 mg capsules
- control group (Placebo Comparator): 21 patients will receive placepo one hour before induction.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gabapentin 600 mg capsules — 21 patients will receive 600 mg oral gabapentin one hour before induction.
  Arms: Gabapentin 600 mg group
Drug: Gabapentin 400 mg capsules — 21 patients will receive 400 mg oral gabapentin one hour before induction.
  Arms: Gabapentin 400 mg group
Drug: Placebo — 21 patients will receive placepo one hour before induction.
  Arms: control group

SUMMARY:
Emergence agitation is a postanesthetic phenomenon that develops in the early phase of recovery from general anesthesia, and is characterized by agitation, disorientation, confusion, and possible violent behavior. Emergence agitation can cause serious events such as self-extubation, bleeding, catheter removal and even falling out of the bed leading to severe injuries . Furthermore, it may lead to injuries to health care providers and increase the demand on human resources.

While its pathogenesis remains unclear, previous studies reported that ENT (ear, nose, and throat) surgical procedures have a higher incidence of emergence agitation in both adults and children.

Emergence agitation is a common phenomenon occurring in 22.2% in adult patients undergoing general anesthesia for nasal surgery .

Gabapentin, agamma-aminobutyricacidanalog, binds the voltage-gated calcium channels of the dorsal root ganglion, at α2-δ subunite. Gabapentin binding to these channels reduces the release of excitatory neurotransmitters preventing the propagation of painful stimuli which makes its use helpful in treatment of postoperative pain and agitation with less side effects compared with benzodiazepines and opioids . Gabapentin has been used in controlling acute perioperative conditions like preoperative anxiety, intraoperative attenuation of hemodynamic response to noxious stimuli and post operative pain, delirium and nausea and vomiting.

A previous study examined the effect of oral gabapentin 600 mg in reducing emergence agitation in adult patients undergowing rhinoplasty, but this study will examine the effect of two different doses of oral gabapentin 400 mg and 600 mg in reducing emergence agitation after nasal surgery.

ELIGIBILITY:
Inclusion Criteria:

* All patients (male/female, American Society of Anesthesiologists physical status I-II, age: 18-60 years) undergoing elective nasal surgery will be eligible for the study.

Exclusion Criteria:

1. hypersensitivity to gabapentin
2. patient refusal
3. epilepsy
4. neurological or psychological conditions that impair communication.
5. current use of gabapentin, psychotropic or opioids medications.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Asessment of emergence agitation | through study completion, an average of 1 year
  Asessment of emergence agitation by Richmond Agitation Sedation Scale(RASS) (score +1 or more) maximum value is +4 (combative) andminimum value is - (unarousable)

SECONDARY OUTCOMES:
Duration of emergence | through study completion, an average of 1 year
  The time in minutes from the discontinuation of anesthesia till the time of spontaneous eye opening or to verbal command
Duration of Post Anesthesia Care Unit (PACU)stay | through study completion, an average of 1 year
  the time in minutes from arrival to Post Anesthesia Care Unit (PACU) to discharge to ward
Number of patients had Postoperative pain | through study completion, an average of 1 year
  Postoperative pain through Numerical Rating Scale (0 represents no pain and 10 represents worst possible pain)
Number of patients required postoperative opioids and total dose. | through study completion, an average of 1 year
Number of patients had postoperative nausea and vomiting (PONV). | through study completion, an average of 1 year
1. Heart rate | through study completion, an average of 1 year
  heart rate in beat per minute (bpm) will be recorded every 5 minutes till the end of operation.
systolic, diastolic and mean arterial blood pressure | through study completion, an average of 1 year
  systolic, diastolic and mean arterial blood pressure in millimeter of mercury (mmHg) will be recorded every 5 minutes till the end of operation.
Oxygen saturation | through study completion, an average of 1 year
  Oxygen saturation in percentage will be recorded every 5 minutes till the end of operation.
Duration of extubation | through study completion, an average of 1 year
  the time in minutes from discontinuation of the anesthetic to removal of endotracheal tube

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Elainy Hospital , Cairo University, Cairo, Cairo Governorate, Egypt

REFERENCES:
- [Background] Badawy AA, Kasem SA, Rashwan D, Al Menesy T, Adel G, Mokhtar AM, Badawy YA. The role of Gabapentin oral solution in decreasing desflurane associated emergence agitation and delirium in children after stabismus surgery, a prospective randomized double-blind study. BMC Anesthesiol. 2018 Jun 20;18(1):73. doi: 10.1186/s12871-018-0533-5. PMID 29925328